CLINICAL TRIAL: NCT02798952
Title: Persistence of Hepatitis B Antibodies, Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Hepatitis B Vaccine, Engerix™-B Kinder (SKF103860) Challenge Dose, in Adolescents Vaccinated With Four Doses of Infanrix™ Hexa (SB217744) During Infancy
Brief Title: A Study to Evaluate Persistence of Hepatitis B Antibodies, Immunogenicity and Safety of Engerix™-B Kinder Challenge Dose, in Adolescents Vaccinated With Four Doses of Infanrix™ Hexa During Infancy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 106794; 2015-003391-74 (EudraCT Number)
Record Dates: First submitted 2016-06-09; First posted 2016-06-14 (Estimated); Results first posted 2019-02-01 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Hepatitis B
Keywords: Hepatitis B antibodies; Safety; Challenge dose; Persistence; Engerix B Kinder; Infanrix hexa; Immunogenicity; Adolescents
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HBV Group (Experimental): Subjects received a single challenge dose of Engerix-B Kinder.
  Interventions: Biological: Engerix-B Kinder

INTERVENTIONS:
Biological: Engerix-B Kinder — Subjects previously primed and boosted with 4 doses of Infanrix hexa vaccine in the first 2 years of life received a single dose of Engerix-B Kinder vaccine as an intramuscular (IM) injection into the deltoid region of the non-dominant arm at 14-15 years of age.

SUMMARY:
The purpose of this study is to assess the long-term persistence of immunity to hepatitis B in adolescents aged 14-15 years who were vaccinated with four doses of Infanrix™-Hexa in the first two years of life and to assess the anamnestic response, immunogenicity, safety and reactogenicity of a single challenge dose of the hepatitis B vaccine Engerix™-B Kinder.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject prior to performance of any study specific procedure.
* In addition to the informed consent that will be signed by the parents/LAR(s), written informed assent of the subject will be sought.
* A male or female between the ages of 14 to 15 at the time of vaccination.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects with documented evidence of previous vaccination with four consecutive doses of Infanrix hexa as part of routine vaccination in Germany: three doses of primary vaccination received by 9 months of age and one booster dose received between 11 and 18 months of age.
* Female subjects of non-childbearing potential may be enrolled in the study.

  * Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy or ovariectomy.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to vaccination, and
  * has a negative pregnancy test on the day of vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the vaccination series.

Exclusion Criteria:

* Child in care.
* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before the dose of study vaccine, or planned use during the study period.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the vaccine dose. For corticosteroids, this will mean prednisone ≥ 0.5 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the dose and ending 30 days after the dose of HBV vaccine administration with the exception of tetanus toxoid, reduced diphtheria toxoid and acellular pertussis vaccine, which can be given as part of routine vaccination practice. Seasonal or pandemic influenza vaccine can be given at any time during the study, and according to the Summary of Product Characteristics and national recommendations.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product (pharmaceutical product or device).
* Evidence of previous hepatitis B booster vaccination since administration of the fourth dose of Infanrix hexa booster in the second year of life.
* History of or intercurrent hepatitis B disease.
* Hepatitis B vaccination at birth.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* Major congenital defects or serious chronic illness including thrombocytopenia and bleeding disorders.
* History of any neurological disorders or seizures.
* Acute disease and/or fever at the time of enrolment.

  * Fever is defined as temperature ≥37.5°C for oral, axillary or tympanic route, or ≥38.0°C for rectal route.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Administration of immunoglobulins and/or any blood products during the period starting 3 months before the dose of study vaccine or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.

Ages: 14 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 302 (Actual)
Dates: Start 2016-08-23 (Actual); Primary Completion 2017-07-05 (Actual); Study Completion 2017-07-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- Germany (14):
  - GSK Investigational Site, Kehl, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Stuttgart, Baden-Wurttemberg
  - GSK Investigational Site, Tuttlingen, Baden-Wurttemberg
  - GSK Investigational Site, Bindlach, Bavaria
  - GSK Investigational Site, Cham, Bavaria
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Frankenthal, Rhineland-Palatinate
  - GSK Investigational Site, Wurzen, Saxony
  - GSK Investigational Site, Berlin
  - GSK Investigational Site, Bramsche
  - GSK Investigational Site, Mönchengladbach
  - GSK Investigational Site, Neumünster

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below)
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=16045

REFERENCES:
- [Background] Schwarz TF, Behre U, Adelt T, Donner M, Suryakiran PV, Janssens W, Mesaros N, Panzer F. Long-term antibody persistence against hepatitis B in adolescents 14-15-years of age vaccinated with 4 doses of hexavalent DTPa-HBV-IPV/Hib vaccine in infancy. Hum Vaccin Immunother. 2019;15(1):235-241. doi: 10.1080/21645515.2018.1509658. Epub 2018 Sep 11. PMID 30118633

RESULTS

PARTICIPANT FLOW:
Groups:
- Engerix-B Kinder Group: Subjects, who were previously primed and boosted with four doses of Infanrix hexa in the first two years of life, received a single challenge dose of Engerix-B Kinder.
Period: Overall Study
Arm/Group | Engerix-B Kinder Group
Started | 302
Completed | 302
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.4 (0.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142
  Male | 160
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - South East Asian Heritage | 1
  Other | 1
  Asian - Central/South Asian Heritage | 1
  White - Caucasian / European Heritage | 293
  African Heritage / African American | 2
  White - Arabic / North African Heritage | 4

OUTCOME MEASURES:

1. Primary Outcome: Anti-Hepatitis B Surface (Anti-HBs) Antibody Concentrations
Description: Concentrations were expressed in geometric mean concentrations (GMCs).
Time Frame: At Day 30.
Population: The analysis was based on the According-to-Protocol cohort for analyses of immunogenicity, which included all subjects who met the eligibility criteria, who complied with the procedures and intervals defined in the protocol and for whom post-vaccination immunogenicity results were available.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 268
mIU/mL | 1975.7 [1436.1 to 2718.1]

2. Secondary Outcome: Anti-HBs Antibody Concentrations
Description: Concentrations were expressed in geometric mean concentrations (GMCs).
Time Frame: At Day 0
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 268
mIU/mL | 15.6 [12.8 to 19.1]

3. Secondary Outcome: Number of Seropositive Subjects for Anti-HBs.
Description: A seropositve subject was defined as a subject with anti-HBs antibody concentrations above the assay cut-off (≥ 6.2 mIU/ml).
Time Frame: At Day 0 and Day 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 268
Participants
  At Day 0 | 163
  At Day 30 | 255

4. Secondary Outcome: Number of Seroprotected Subjects for Anti-HBs.
Description: A seroprotected subject was defined as a subject with anti-HBs antibody concentrations equal to or above 10 milli-International units per milliliter (mIU/ml).
Time Frame: At Day 0 and day 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 268
Participants
  At Day 0 | 144
  At Day 30 | 250

5. Secondary Outcome: Number of Subjects With Anti-HBs Concentrations Above the Cut-off.
Description: The cut-off of the assay was ≥ 100 mIU/mL.
Time Frame: At Day 0 and Day 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 268
Participants
  At Day 0 | 45
  At Day 30 | 234

6. Secondary Outcome: Number of Subjects With an Anamnestic Response to the Hepatitis B Challenge Dose.
Description: Anamnestic response was defined as:
  For initially seronegative subjects: antibody concentration ≥10mIU/mL. For initially seropositive subjects: antibody concentration at least four times the pre-challenge antibody concentration.
Time Frame: At Day 30
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 268
Participants | 248

7. Secondary Outcome: Number of Subjects With Any Solicited Local and General Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling at injection site. Solicited general symptoms assessed were fatigue, gastrointestinal symptoms, headache and fever (defined as axillary temperature ≥ 37.5°C).
Time Frame: Within 4 days (Day 0 - Day 3) after the vaccination
Population: The analysis was based on the Total Vaccinated cohort, which included all subjects who received the study vaccine and had their symptoms sheet completed .
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 301
Participants
  Redness | 65
  Pain | 101
  Swelling | 32
  Fatigue | 91
  Gastrointestinal symptoms | 33
  Headache | 76
  Fever | 16

8. Secondary Outcome: Number of Subjects With Unsolicited Adverse Events (AEs)
Description: An unsolicited AE was defined as any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Within 31 days (Day 0 - Day 30) after the vaccination.
Population: The analysis was based on the Total Vaccinated cohort, which included all subjects who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 302
Participants | 55

9. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs)
Description: An SAE was defined as any untoward medical occurrence that: resulted in death, was life-threatening, required hospitalization or prolongation of existing hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 0 to Day 30
Population: The analysis was based on the Total Vaccinated cohort, which included all subjects who received the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Engerix-B Kinder Group
Number analyzed (Participants) | 302
Participants | 2

ADVERSE EVENTS:
Time Frame: Solicited local and general symptoms: during the 4-day (Day 0-3) follow-up period after vaccination. Unsolicited AE(s) and SAE(s): during the entire study period (Days 0-30).
Arm/Group | Engerix-B Kinder Group
All-Cause Mortality (participants affected / at risk) | 0/302
Serious Adverse Events (participants affected / at risk) | 2/302
Other Adverse Events (participants affected / at risk) | 197/302
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engerix-B Kinder Group (N=302)
Meniscus injury (Injury, poisoning and procedural complications) | 1 (1)
Eating disorder (Psychiatric disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engerix-B Kinder Group (N=302)
Fatigue (General disorders) | 91 (91)
Gastrointestinal disorder (Gastrointestinal disorders) | 33 (33)
Headache (Nervous system disorders) | 79 (80)
Injection site erythema (General disorders) | 65 (65)
Injection site pain (General disorders) | 101 (101)
Injection site swelling (General disorders) | 32 (32)
Pyrexia (General disorders) | 16 (16)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT02798952/SAP_000.pdf
  • Study Protocol (2015-11-06): https://cdn.clinicaltrials.gov/large-docs/52/NCT02798952/Prot_001.pdf